CLINICAL TRIAL: NCT01646034
Title: High-dose Alkylating Chemotherapy in Oligo-metastatic Breast Cancer Harboring Homologous Recombination Deficiency
Brief Title: High Dose Chemotherapy in Oligo-metastatic Homologous Recombination Deficient Breast Cancer
Acronym: Oligo
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N12OLG; 2012-000838-19 (EudraCT Number)
Record Dates: First submitted 2012-06-14; First posted 2012-07-20 (Estimated); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer
Keywords: oligo metastatic; HRD deficiency
MeSH Terms: conditions — Breast Neoplasms | interventions — Carboplatin; Thiotepa; Cyclophosphamide; Drug Therapy; Docetaxel; Doxorubicin; Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intensified alkylating chemotherapy (Experimental): a course chemotherapy with high dose cyclophosphamide, G-CSF and peripheral blood progenitor cell (PBPC) harvest followed by tandem intermediate-dose alkylating therapy (miniCTC, carboplatin 800 mg/m2, thiotepa 240 mg/m2, and cyclophosphamide 3000 mg/m2) with PBPC-reinfusion.
  Interventions: Drug: carboplatin, thiotepa, and cyclophosphamide
- three cycles of chemotherapy (Active Comparator): three cycles of chemotherapy depending on previously received agents
  chemotherapy naïve;three cycles of docetaxel, doxorubicin, and cyclophosphamide previously received anthracyclines without taxanes;three cycles of carboplatin and paclitaxel previously received anthracyclines and taxanes;three cycles of carboplatin and gemcitabine
  Interventions: Drug: chemotherapy (docetaxel, doxorubicin, cyclofosfamide, carboplatin, paclitaxel, gemcitabine)

INTERVENTIONS:
Drug: carboplatin, thiotepa, and cyclophosphamide — tandem intermediate-dose alkylating therapy: carboplatin 800 mg/m2, thiotepa 240 mg/m2, and cyclophosphamide 3000 mg/m2) with PBPC-reinfusion.
  Arms: intensified alkylating chemotherapy
Drug: chemotherapy (docetaxel, doxorubicin, cyclofosfamide, carboplatin, paclitaxel, gemcitabine) — * chemotherapy naïve;three cycles of docetaxel, doxorubicin, and cyclofosfamide
  * chemotherapy naïve;1 cycle of dose-dense Adriamycin and cyclophosphamide followed by 4 cycles of carboplatin and paclitaxel
  * previously received anthracyclines without taxanes;three cycles of carboplatin and paclitaxel
  * previously received anthracyclines and taxanes;three cycles of carboplatin and gemcitabine
  Arms: three cycles of chemotherapy

SUMMARY:
This study investigates the effect of high-dose alkylating chemotherapy compared with standard chemotherapy as part of a multimodality treatment approach in patients with oligo-metastatic breast cancer harboring homologous recombination deficiency.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed infiltrating breast cancer
2. Oligometastatic disease defined as one to three distant metastatic lesions, with or without primary tumor, local recurrence, or locoregional lymph node metastases, including the ipsilateral axillary, parasternal, and periclavicular regions. All lesions must be amenable to resection or radiotherapy with curative intent. Staging examinations must have included a PET-CT-scan and a MRI of the liver in case of liver metastases. Clustered lymph nodes that can be irradiated with curative intent in a single field are defined as a single lesion. Histologic or cytologic confirmation of at least one distant metastatic lesion is required.
3. No prior line of chemotherapy for metastatic disease (a maximum of 3 months of palliative endocrine therapy is allowed).
4. The tumor must be HER2-negative (either score 0 or 1 at immunohistochemistry or negative at in situ hybridization in case of score 2 or 3 at immunohistochemistry).
5. The tumor is deficient in homologous recombination and/or the patient has a deleterious germline BRCA1 or BRCA2 mutation.
6. At least stable disease of all tumor lesions after three courses of induction chemotherapy
7. Age ≥18 years
8. World Health Organisation (WHO) performance status 0 or 1
9. Adequate bone marrow function (ANC ≥1.0 x 109/l, platelets ≥100 x 109/l)
10. Adequate hepatic function (ALAT, ASAT and bilirubin ≤2.5 times upper limit of normal)
11. Adequate renal function (creatinine clearance ≥60 ml/min)
12. If clinically recommended echocardiography, MUGA, or MRI to evaluate if LVEF ≥50%;
13. Signed written informed consent
14. Able to comply with the protocol

Exclusion Criteria:

* No malignancy other than breast cancer, unless treated with curative intent without the use of chemotherapy or radiation therapy
* No current pregnancy or breastfeeding. Women of childbearing potential must use adequate contraceptive protection.
* No concurrent anti-cancer treatment or investigational drugs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2014-09; Primary Completion 2023-01 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Event free survival | assessed up to 120 months
  time from randomization to local recurrence, second primary, distant recurrence or death, whichever comes first

SECONDARY OUTCOMES:
Difference in median overall survival | assessed up to 120 months
  time from randomization to death from any cause
Difference in percentage of patients with grade >2 hematologic toxicity (CTCAE v4.0) | 6 months after start of treament
  Difference in percentage of patients with grade >2 hematologic toxicity (CTCAE v4.0)
Difference in percentage of patients with grade >2 non-hematologic toxicity (CTCAE v4.0) | 6 months after start of treatment
  Difference in percentage of patients with grade >2 non-hematologic toxicity (CTCAE v4.0)
Difference in quality of life (EORTC QLQ-C30 v 3.0) | 6 and 12 months post treatment
  Difference in quality of life (EORTC QLQ-C30 v 3.0)
Difference in event free survival | assessed up to 120 months
  o Difference in event free survival in the subgroups based on:
  * Estrogen receptor status;
  * Origin of the oligo-metastatic lesion (lymphnodes versus bone versus visceral metastases);
  * Primary or recurrent oligometastatic breast cancer;
  * BRCA1 mutation/profile or BRCA2 mutation/profile;
  * HRD based on BRCA1 or BRCA2 mutation and HRD based on BRCA1-like and/or BRCA2-like profile.

CONTACTS AND LOCATIONS:
Overall Officials: Gabe S Sonke, MD, Principal Investigator — NKI-AVL, Amsterdam
Locations (1):
- NKI-AVL, Amsterdam, Netherlands

REFERENCES:
- [Derived] van Ommen-Nijhof A, Steenbruggen TG, Wiersma TG, Balduzzi S, Daletzakis A, Holtkamp MJ, Delfos M, Schot M, Beelen K, Siemerink EJM, Heijns J, Mandjes IA, Wesseling J, Rosenberg EH, Vrancken Peeters MJT, Linn SC, Sonke GS. Intensified alkylating chemotherapy for patients with oligometastatic breast cancer harboring homologous recombination deficiency: Primary outcomes from the randomized phase III OLIGO study. Eur J Cancer. 2024 Dec;213:115083. doi: 10.1016/j.ejca.2024.115083. Epub 2024 Oct 20. PMID 39489924